CLINICAL TRIAL: NCT01107301
Title: Vascular Consequences of ADHD Medication Use in Children and Adolescents
Brief Title: Vascular Effects of Attention Deficit Hyperactivity Disorder (ADHD) Medications in Youth
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0912M74832
Record Dates: First submitted 2010-04-07; First posted 2010-04-20 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: ADHD
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
4.4 million children and adolescents in the United States have been diagnosed with attention deficit hyperactivity disorder (ADHD) and more than half are treated with medication. Most ADHD medications are stimulants, which activate the sympathetic nervous system (SNS). SNS activation is closely associated with vascular functional and mechanical abnormalities. Therefore, ADHD medications, via instigating SNS activation and altering the hemodynamic profile, may have untoward effects on the vasculature and increase risk of developing cardiovascular disease in children and adolescents who use them.

Our overall objective in this study is to determine whether ADHD medication use is associated SNS activation, endothelial dysfunction, and arterial stiffness in children and adolescents. We will address this objective by conducting a case-control study and obtain non-invasive measures of SNS activation, endothelial function, and arterial stiffness in children and adolescents (8-17 years old) with (using stimulant medication) and without ADHD.

DETAILED DESCRIPTION:
SPECIFIC AIMS AND HYPOTHESES

Our overall objective in this study is to determine whether ADHD medication use is associated SNS activation, endothelial dysfunction, and arterial stiffness in children and adolescents.

Our hypothesis is:

Children and adolescents taking ADHD medications will have higher SNS activation, lower digital reactive hyperemia, and higher pulse wave velocity and aortic augmentation index compared to sibling controls without ADHD.

Study Design We will obtain non-invasive measures of SNS activation (heart rate variability), endothelial function (digital reactive hyperemia and brachial artery flow-mediated dilation), and arterial stiffness (carotid-radial pulse wave velocity; aortic augmentation index) in youth taking ADHD stimulant medication and in their healthy siblings without ADHD.

Study visits will be conducted at the Clinical and Translational Science Institute (CTSI) at the University of Minnesota. All vascular testing will occur in the Vascular Biology Laboratory within the CTSI.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years old
* Current use of ADHD stimulant drug therapy limited to methylphenidates or amphetamines
* Sibling without ADHD between the ages of 6-18 years old

Exclusion Criteria:

• Known (diagnosed) cardiac disease

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Eighty youth who are taking ADHD stimulant medication and eighty of their healthy siblings without ADHD.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | Baseline
  Carotid-radial pulse wave velocity and aortic augmentation index.

SECONDARY OUTCOMES:
SNS activation | Baseline
  Heart rate variability.
Endothelial Function | Baseline
  Digital reactive hyperemia and brachial artery flow-mediated dilation

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States